CLINICAL TRIAL: NCT04382664
Title: Efficacy and Safety of UV1 Vaccination in Combination With Nivolumab and Ipilimumab as First Line Treatment of Patients With Unresectable or Metastatic Melanoma (INITIUM Study)
Brief Title: UV1 Vaccination Plus Nivolumab and Ipilimumab in Treatment of Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultimovacs ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UV1-202
Record Dates: First submitted 2020-04-27; First posted 2020-05-11 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — sargramostim; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UV1 vaccination + nivolumab and ipilimumab (Experimental): UV1 vaccination + nivolumab and ipilimumab
  Interventions: Biological: UV1; Biological: Sargramostim; Biological: Ipilimumab; Biological: Nivolumab
- Nivolumab and ipilimumab (Active Comparator): Nivolumab and ipilimumab
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: UV1 — UV1 vaccine (300 μg) will be injected intradermally.
  Arms: UV1 vaccination + nivolumab and ipilimumab
Biological: Sargramostim — Sargramostim (75 μg) is used as a vaccine adjuvant.
  Other Names: Leukine
  Arms: UV1 vaccination + nivolumab and ipilimumab
Biological: Ipilimumab — Ipilimumab is dosed according to label.
  Other Names: Yervoy
Biological: Nivolumab — Nivolumab is dosed according to label.
  Other Names: Opdivo

SUMMARY:
This is a randomized, open label study to investigate efficacy and safety of UV1 vaccination in combination with nivolumab and ipilimumab as first line treatment of adult patients with histologically confirmed unresectable metastatic melanoma.

DETAILED DESCRIPTION:
This is a randomized, open label study to investigate efficacy and safety of UV1 vaccination in combination with nivolumab and ipilimumab as first line treatment of adult patients with histologically confirmed unresectable metastatic melanoma.

Patients in the experimental arm will receive 8 UV1 vaccinations over 4 cycles of nivolumab and ipilimumab. Patients in the control arm will receive 4 cycles of nivolumab and ipilimumab. Patients in both arms will start maintenance therapy 6 weeks after the last dose of induction therapy, nivolumab at a dose of 480 mg every 4 weeks.

All patients will be followed up until death or until the end of the study.

To support the Extended Exploratory Cohort of the study, an additional 20 patients at selected sites will be enrolled in a single arm UV1 cohort for collection of additional biological material. These patients are in addition to the 156 randomized patients in the main part of the study and will not be included in the main analysis of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years of age at the time of signing the ICF.
2. Histologically confirmed diagnosis of unresectable stage IIIB D, or unresectable stage IV malignant melanoma.
3. Eligible for combination treatment with nivolumab and ipilimumab.
4. An ECOG performance status of 0 or 1.
5. Adequate organ function as indicated by the following laboratory values:

   Hematological
   1. Absolute neutrophil count ≥1,500/µL
   2. Platelet count ≥100 x 103/µL
   3. Hemoglobin ≥9 g/dL or ≥5.6 mmol/L Renal
   4. Creatinine ≤1.5 x upper limit of normal (ULN) Hepatic
   5. Total bilirubin ≤1.5 x ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 ULN
   6. Aspartate aminotransferase/serum glutamic oxaloacetic transaminase and alanine aminotransferase/serum glutamic pyruvic transaminase ≤2.5 x ULN for patients without liver metastasis or ≤5 x ULN for patients with liver metastasis.
6. Male patients who are sexually active with a female of childbearing potential must agree to use an adequate method of contraception.
7. Women of childbearing potential (WOCBP) must have a negative urine or serum/plasma pregnancy test.
8. WOCBP must use adequate contraception.

Exclusion Criteria:

1. Previous non melanoma malignancies unless curatively treated and complete remission was achieved at least 2 years prior to randomization. Patients with prior curatively treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or carcinoma in situ of the breast, or other in situ cancers are allowed irrespective of time passed since curative treatment. Patients with prior completely resected malignant melanoma are also allowed.
2. Known brain metastases or leptomeningeal metastases. If a patient experiences neurological symptoms indicative of brain metastases, a brain MRI should be performed.
3. Diagnosis of uveal or ocular melanoma.
4. Known history or any evidence of active, non-infectious pneumonitis.
5. History of New York Heart Association class 3-4 congestive heart failure or history of myocardial infarction within 6 months of starting induction therapy.
6. Active infection requiring systemic treatment.
7. Diagnosis of immunodeficiency.
8. Known history of severe hypersensitivity reactions to nivolumab, ipilimumab, sargramostim, or their excipients.
9. Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
10. History of or active hepatitis B (hepatitis B surface antigen reactive) or active hepatitis C (hepatitis C virus antibody).
11. Women who are breastfeeding.
12. Prior systemic treatment for unresectable stage IIIB D or unresectable stage IV malignant melanoma.
13. Systemic corticosteroid treatment (doses exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive treatment within 7 days prior to the first dose of induction therapy.
14. Receipt of a live vaccine within 30 days prior to start of induction therapy.
15. Receipt of any other investigational treatment within 4 weeks of the first dose of induction therapy.
16. Any medical, psychological, or social condition that would make it difficult for the patient to participate in the study and comply with the study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Lewis, Principal Investigator — University of Colorado Hospital - Anschutz Cancer Pavilion
Locations (37):
- United States (20):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of California Irvine Health, Orange, California
  - California Cancer Associates for Research & Excellence (CCARE, San Marcos, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Saint John's Health Center - John Wayne Cancer Institute (JWCI), Santa Monica, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Holy Cross Medical Group, Fort Lauderdale, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Rush University Medical Center - Rush University Cancer Center, Chicago, Illinois
  - NorthShore University Research Institute, Evanston, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Nebraska Cancer Specialists- Midwest Cancer Center, Papillion, Nebraska
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - State University of New York (SUNY) Upstate Medical University, New York, New York
  - University of Rochester, Rochester, New York
  - NorthShore University HealthSystem, Greenville, South Carolina
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
- Belgium (4):
  - Antwerp University Hospital, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Leuven University Hospital, Leuven
  - GZA Hospital Sint-Augustinus, Wilrijk
- Norway (7):
  - Ålesund Hospital- Helse Sunnmore HF, Ålesund
  - Sykehuset Østfold HF, Grålum
  - Sørlandet Sykehus HF(SSHF), Kristiansand
  - Oslo University Hospital - The Norwegian Radium Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - Universitetssykehuset Nord-Norge HF, Tromsø
  - St. Olavs Hospital HF, Trondheim
- United Kingdom (6):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology and Oncology Centre, Bristol
  - Velindre NHS Trust, Cardiff
  - The Royal Free London NHS Foundation Trust - The Royal Free Hospital, London
  - Royal Marsden Hospital - Institute of Cancer Research - Chelsea, London
  - Cancer Research UK Manchester Institute, Manchester
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford

RESULTS

PARTICIPANT FLOW:
Groups:
- UV1 Vaccination + Nivolumab and Ipilimumab: UV1 vaccination + nivolumab and ipilimumab
  UV1 vaccination includes sargramostim (75 μg), used as a vaccine adjuvant, and the UV1 vaccine (300 μg). Both injected intradermally.
  Ipilimumab: Ipilimumab is dosed according to label.
  Nivolumab: Nivolumab is dosed according to label.
Period: Overall Study
Arm/Group | UV1 Vaccination + Nivolumab and Ipilimumab | Nivolumab and Ipilimumab
Started | 78 | 78
Completed | 75 | 76
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UV1 Vaccination + Nivolumab and Ipilimumab | Nivolumab and Ipilimumab | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 55 | 95
  >=65 years | 38 | 23 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 53 | 49 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 75 | 76 | 151
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Belgium | 17 | 11 | 28
  United States | 29 | 34 | 63
  Norway | 11 | 16 | 27
  United Kingdom | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: PFS Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (by Blinded Independent Central Review (BICR)
Description: Compare progression free survival (PFS) of UV1 vaccination in combination with nivolumab and ipilimumab to that of nivolumab and ipilimumab
Time Frame: Time from randomization to progressive disease (PD) or death from any cause (approximately 44 months)
Population: Intention To Treat population (IIT)
Measure: Count of Participants; unit: Participants
Arm/Group | UV1 Vaccination + Nivolumab and Ipilimumab | Nivolumab and Ipilimumab
Number analyzed (Participants) | 78 | 78
Participants | 35 | 34
Statistical Analysis 1: Comparison: UV1 Vaccination + Nivolumab and Ipilimumab vs Nivolumab and Ipilimumab; Test type: Superiority; p = 0.845, Regression, Cox; Hazard Ratio (HR) = 0.95, 80% CI 2-sided [0.694 to 1.309]

2. Secondary Outcome: Overall Survival
Description: Compare Overall Survival of UV1 vaccination in combination with nivolumab and ipilimumab to that of nivolumab and ipilimumab .
Time Frame: Time from randomization to death from any cause /follow-up until 70 PFS events/18 months post rand, approximately 44 months.
Reporting Status: Not Posted

3. Secondary Outcome: ORR Per RECIST 1.1
Description: Compare the objective response rate (ORR) of UV1 vaccination in combination with nivolumab and ipilimumab to that of nivolumab and ipilimumab.
Time Frame: Number of complete and partial responses during the study, approximately 44 months.
Reporting Status: Not Posted

4. Secondary Outcome: DOR Per RECIST 1.1
Description: Compare duration of response (DOR) of UV1 vaccination in combination with nivolumab and ipilimumab to that of nivolumab and ipilimumab.
Time Frame: Time from first CR or PR to PD or death from any cause, approximately 44 months.
Reporting Status: Not Posted

5. Secondary Outcome: Evaluation of Adverse Events, Vital Signs, Laboratory Assessments and ECOG Performance Status
Description: Compare the safety of UV1 vaccination in combination with nivolumab and ipilimumab to that of nivolumab and ipilimumab. Safety will be listed and summarized descriptively by treatment arm comparing number of participants with observation and changes from baseline and at each visit related to AEs, deaths, vital signs (weight (kg), systolic and diastolic blood pressure (mmHg), pulse rate (bpm), body temperature (°C)), laboratory assessments and ECOG performance status (Grade 0 - Grade 5).
Time Frame: Time from randomization to end of study, approximately 47 months.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Immunological Mechanisms
Description: To elucidate the immunological mechanisms underlying the interplay between immune activation provoked by UV1 vaccination and inhibition of tumor resistance mechanisms and peripheral immune tolerance induced by checkpoint blockade and how biological factors affect the efficacy of the combination therapy. This will be evaluated by change in immune- and tumor-related gene, cell, and protein profiles in blood over time in both treatment arms (analysis of plasma proteins, cell-free plasma DNA, and cellular genomic DNA).
Time Frame: Time from randomization to end of study to readout of primary objectives, approximately 44 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 44 months
Arm/Group | UV1 Vaccination + Nivolumab and Ipilimumab | Nivolumab and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 22/76 | 17/78
Serious Adverse Events (participants affected / at risk) | 40/76 | 43/78
Other Adverse Events (participants affected / at risk) | 76/76 | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UV1 Vaccination + Nivolumab and Ipilimumab (N=76) | Nivolumab and Ipilimumab (N=78)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Myocarditis (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 3
Adrenal insufficiency (Endocrine disorders) | 2 | 1
Immune-mediated thyroiditis (Endocrine disorders) | 0 | 2
Addisons disease (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 4 | 7
Immune-mediated enterocolitis (Gastrointestinal disorders) | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Enteritis (Gastrointestinal disorders) | 1 | 1
Immune-mediated pancreatitis (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 0
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 4 | 3
Hepatitis (Hepatobiliary disorders) | 1 | 4
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0
Anaphylactic shock (Immune system disorders) | 1 | 1
Contrast media reaction (Immune system disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1
Infusion related reaction (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
COVID-19 (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 1
Meningitis aseptic (Infections and infestations) | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Respiratory rate increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UV1 Vaccination + Nivolumab and Ipilimumab (N=76) | Nivolumab and Ipilimumab (N=78)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Cardiac disorders (Cardiac disorders) | 8 | 5
Hyperthyroidism (Endocrine disorders) | 11 | 8
Hypothyroidism (Endocrine disorders) | 9 | 10
Hypophysitis (Endocrine disorders) | 2 | 9
Adrenal insufficiency (Endocrine disorders) | 4 | 3
Vision blurred (Eye disorders) | 2 | 5
rfw (Gastrointestinal disorders) | 26 | 21
Diarrhoea (Gastrointestinal disorders) | 24 | 22
Vomiting (Gastrointestinal disorders) | 13 | 13
Constipation (Gastrointestinal disorders) | 11 | 8
Colitis (Gastrointestinal disorders) | 5 | 12
Abdominal pain (Gastrointestinal disorders) | 8 | 5
Immune-mediated enterocolitis (Gastrointestinal disorders) | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 31 | 33
Pyrexia (General disorders) | 21 | 10
Injection site erythema (General disorders) | 13 | 0
Injection site reaction (General disorders) | 11 | 0
Oedema peripheral (General disorders) | 7 | 4
Chills (General disorders) | 4 | 5
Influenza like illness (General disorders) | 4 | 1
Injection site pain (General disorders) | 4 | 0
Vaccination site hyperaesthesia (General disorders) | 4 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 6 | 8
Hepatitis (Hepatobiliary disorders) | 4 | 5
Infusion related reaction (Immune system disorders) | 6 | 4
COVID-19 (Infections and infestations) | 4 | 5
Oral candidiasis (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 5 | 1
Alanine aminotransferase increased (Investigations) | 11 | 15
Aspartate aminotransferase increased (Investigations) | 11 | 13
Blood creatinine increased (Investigations) | 3 | 7
Weight decreased (Investigations) | 4 | 5
Blood alkaline phosphatase increased (Investigations) | 3 | 4
Blood bilirubin increased (Investigations) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 15 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2
Headache (Nervous system disorders) | 9 | 15
Insomnia (Psychiatric disorders) | 4 | 4
Renal and urinary disorders (Renal and urinary disorders) | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 21
Rash (Skin and subcutaneous tissue disorders) | 19 | 23
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 4
Hypertension (Vascular disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT04382664/Prot_SAP_000.pdf